CLINICAL TRIAL: NCT00845156
Title: Alpha Lipoic Acid and Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H6820-30422
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Insulin Resistance
Keywords: Diabetes; Insulin resistance; healthy controls; anti oxidants
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anti-Oxidant (Active Comparator): Alpha Lipoic Acid
  Interventions: Dietary Supplement: Alpha Lipoic Acid
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Alpha Lipoic Acid

INTERVENTIONS:
Dietary Supplement: Alpha Lipoic Acid — Two 400 mg tablets of Alpha Lipic Acid are taken 3 times daily

SUMMARY:
Subjects will be screened with a 2 hour oral glucose tolerance test. After this screening visit, their insulin resistance will be measured. Subjects will then be given either alpha lipoic acid (antioxidant) or placebo for 6 weeks. The insulin resistance test will be repeated after the 6 weeks. We believe these studies will confirm the beneficial effect of alpha lipoic acid on insulin sensitivity.

DETAILED DESCRIPTION:
We propose to perform a placebo-controlled study of Alpha Lipoic Acid (LA) administration in a cohort of non-obese, non-diabetic, insulin resistant subjects. The insulin sensitivity of 180 subjects will be initially estimated by measuring fasting glucose and insulin levels (homeostasis model assessment) and oral glucose tolerance test (OGTT). The 60 most insulin resistant subjects will then be randomized to 6 weeks of therapy with either 600 mg three times a day of LA or placebo. To quantitate the ALA-induced improvements, euglycemic hyperinsulinemic clamps to evaluate insulin sensitivity, OGTT using deuterated glucose to evaluate glycolytic glucose disposal, and muscle biopsies to evaluate insulin signaling pathways, will be performed before and after treatment. We believe these studies will (1) confirm the beneficial effect of CR-ALA on insulin sensitivity; (2) further our understanding of the molecular mechanisms of LA action; and (3) because these insulin resistant subjects are at risk for the development of type 2 diabetes, the Metabolic Syndrome, and coronary artery disease (CAD), a demonstration of the beneficial effects of LA on insulin action could ultimately have important public health consequences.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, not exercising regularly

Exclusion Criteria:

* Diabetes, Impaired glucose tolerance, Heart disease, Liver disease, HIV, abnormal TSH results, other abnormal lab values

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2008-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Insulin Resistance | 0 months and 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Umesh Masharani, MD, Principal Investigator — University of California, San Francisco; Martha Kennedy, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California at San Francisco, San Francisco, California, United States